CLINICAL TRIAL: NCT01944839
Title: A Phase 3 Randomized, Double-masked, Controlled Trial to Establish the Safety and Efficacy of Intravitreous Administration of Fovista® (Anti PDGF-B Pegylated Aptamer) Administered in Combination With Lucentis® Compared to Lucentis® Monotherapy in Subjects With Subfoveal Neovascular Age-related Macular Degeneration.
Brief Title: A Phase 3 Safety and Efficacy Study of Fovista® (E10030) Intravitreous Administration in Combination With Lucentis® Compared to Lucentis® Monotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPH1002
Record Dates: First submitted 2013-09-09; First posted 2013-09-18 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2018-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet AMD; choroidal neovascularization; Fovista®; E10030; Lucentis®
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — E10030 aptamer; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E10030 + ranibizumab (Experimental): E10030 1.5 mg intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  Interventions: Drug: E10030; Drug: ranibizumab
- Sham + ranibizumab (Active Comparator): E10030 sham intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  Interventions: Drug: ranibizumab; Drug: E10030 sham intravitreal injection

INTERVENTIONS:
Drug: E10030
  Other Names: Fovista®
  Arms: E10030 + ranibizumab
Drug: ranibizumab
  Other Names: Lucentis®
Drug: E10030 sham intravitreal injection — Pressure on the eye with a syringe with no needle
  Other Names: Sham
  Arms: Sham + ranibizumab

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of intravitreal administration of Fovista® administered in combination with Lucentis® compared to Lucentis® monotherapy in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to the following dose groups:

* Fovista® 1.5 mg/eye + Lucentis® 0.5 mg/eye
* Fovista® sham + Lucentis® 0.5 mg/eye

Subjects will be treated for a total of 24 months with active Fovista® or sham in combination with Lucentis® with the primary endpoint at 12 months.

Primary Efficacy Endpoint:

The primary efficacy endpoint is the mean change in visual acuity (ETDRS letters) from baseline at the month 12 visit.

Safety Endpoints:

Safety endpoints include adverse events, vital signs, ophthalmic variables [ophthalmic examination, intraocular pressure (IOP), fluorescein angiogram (FA), optical coherence tomography (OCT)], ECG, and laboratory variables.

Approximately 622 subjects will be randomized into one of the two treatment cohorts (311 patients per dose group).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years
* Active subfoveal choroidal neovascularization (CNV) secondary to AMD
* Presence of sub-retinal hyper-reflective material (SD-OCT)

Exclusion Criteria:

* Any prior treatment for AMD in the study eye prior to the Day 1 visit, except oral supplements of vitamins and minerals
* Any prior intravitreal treatment in the study eye prior to the Day 1 visit, regardless of indication (including intravitreal corticosteroids)
* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication
* Subjects with subfoveal scar or subfoveal atrophy are excluded
* Diabetes mellitus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (47):
  - Phoenix, Arizona
  - Bakersfield, California
  - Beverly Hills, California
  - Los Angeles, California
  - San Francisco, California
  - Santa Barbara, California
  - Colorado Springs, Colorado
  - Bridgeport, Connecticut
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Fort Myers, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Marietta, Georgia
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Leawood, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - Jackson, Michigan
  - Southfield, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Portsmouth, New Hampshire
  - Northfield, New Jersey
  - Albuquerque, New Mexico
  - Great Neck, New York
  - Shirley, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Ashland, Oregon
  - Camp Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Ladson, South Carolina
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Madison, Wisconsin
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Belgium (2):
  - Deurne, Antwerpen
  - Leuven, Vlaams-Brabant
- Brazil (4):
  - Goiânia, Goiás
  - Porto Alegre, Rio Grande do Sul
  - Minas Gerais
  - São Paulo
- Canada (10):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Czechia (5):
  - Brno
  - Kralovice
  - Libeň
  - Olomouc
  - Prague
- Estonia (3):
  - Harju
  - Tallinn
  - Tartu
- Italy (9):
  - Ancona
  - Bologna
  - Ferrara
  - Florence
  - Milan
  - Padua
  - Roma
  - Torino
  - Udine
- Riga, Latvia
- Poland (5):
  - Bydgoszcz
  - Katowice
  - Lodz
  - Warsaw
  - Wroclaw
- Slovakia (3):
  - Banská Bystrica
  - Bratislava
  - Trenčín
- Switzerland (4):
  - Basel
  - Bern
  - Lausanne
  - Zurich
- United Kingdom (6):
  - Belfast
  - Liverpool
  - London
  - Plymouth
  - Southampton
  - Surrey Quays

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Groups:
- E10030 + Ranibizumab: E10030 1.5 mg intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  E10030
  ranibizumab
- Sham + Ranibizumab: E10030 sham intravitreal injection + ranibizumab 0.5 mg intravitreal injection
  ranibizumab
  E10030 sham intravitreal injection: Pressure on the eye with a syringe with no needle
Period: Overall Study
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab
Started | 309 | 310
Completed | 287 | 282
Not Completed | 22 | 28
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 10 | 5
Not completed — Withdrawal by Subject | 9 | 17
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject non-compliance | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab | Total
Number analyzed (Participants) | 309 | 310 | 619
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.98) | 76.9 (8.04) | NA (NA) — not calculated
Age, Customized [Count of Participants; unit: Participants]
  Adults 18-64 years | 26 | 20 | 46
  Adults 65 - 84 years | 243 | 233 | 476
  85 years and over | 40 | 57 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 196 | 377
  Male | 128 | 114 | 242
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 106 | 104 | 210
  Czechia | 42 | 42 | 84
  United Kingdom | 13 | 14 | 27
  Switzerland | 3 | 4 | 7
  Canada | 14 | 9 | 23
  Austria | 5 | 5 | 10
  Latvia | 21 | 25 | 46
  Belgium | 1 | 0 | 1
  Poland | 23 | 23 | 46
  Brazil | 8 | 8 | 16
  Italy | 56 | 62 | 118
  Slovakia | 5 | 4 | 9
  Estonia | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity From Baseline to 12 Months
Description: The primary efficacy endpoint is the mean change in visual acuity (ETDRS letters) from baseline to the month 12 visit. Higher ETDRS letters represents higher vision and a higher change in ETDRS letters represents better functioning.
Time Frame: 12 Months
Measure: Mean (Standard Error); unit: letters
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab
Number analyzed (Participants) | 309 | 310
letters | 10.74 (0.86) | 9.82 (0.86)

ADVERSE EVENTS:
Time Frame: Up to 12 months of exposure
Description: The efficacy (ITT) population, defined as all subjects randomized and received at least one dose of study drug, is different than the safety population, where all subjects who have received at least one dose of E10030 are analyzed as on that group. There was one subject who was randomized to Sham+Ranibizumab but was mis-treated with one dose of E10030 and therefore was analyzed in the E10030+ranibizuma group for safety purposes. This is the same explanation for the SAE and Mortality tables.
Arm/Group | E10030 + Ranibizumab | Sham + Ranibizumab
All-Cause Mortality (participants affected / at risk) | 6/310 | 2/309
Serious Adverse Events (participants affected / at risk) | 48/310 | 36/309
Other Adverse Events (participants affected / at risk) | 123/310 | 114/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 + Ranibizumab (N=310) | Sham + Ranibizumab (N=309)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gilioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Device failure (General disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoidal haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oroantral fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric rupture (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Endophthalmitis (Infections and infestations) | 3 (3) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster meningoencephalitis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 + Ranibizumab (N=310) | Sham + Ranibizumab (N=309)
Intraocular pressure increased (Investigations) | 43 (157) | 30 (78)
Conjunctival haemorrhage (Eye disorders) | 60 (197) | 56 (177)
Eye pain (Eye disorders) | 23 (29) | 26 (47)
Punctate keratitis (Eye disorders) | 15 (22) | 18 (30)
Nasopharyngitis (Infections and infestations) | 19 (20) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees not to individually publish the results of the Study without Ophthotech's prior written consent. Institution may participate in a joint, multi-center publication of the Study results with other investigators and/or institutions only, upon the prior written consent of Ophthotech.